CLINICAL TRIAL: NCT02865044
Title: A Randomized, Controlled, Crossover Study to Evaluate the Acute Bioavailability of Eicosapentaenoic Acid andDocosahexaenoic Acid From a DietarySupplement in Healthy Men and Women: A 72-Hour Study With Controlled Feeding
Brief Title: Study to Evaluate the Acute Bioavailability of EPA and DHA From a DietarySupplement in Healthy Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calanus (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO 1505
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Fatty Acids; Fish Oil; Marine Copepod; Fatty Acid Absorption
MeSH Terms: interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wax Ester Marine Oil (Active Comparator): Active: Wax ester marine oil (Calanus oil; 4 g providing 260 mg EPA and 156 mg DHA; 8 capsules)
  Interventions: Other: Wax Ester Marine Oil
- Ethyl Ester Marine Oil (Other): Control: Ethyl ester (EE) marine oil (Lovaza OM3 EE; 1 g providing 465 mg EPA and 375 mg DHA; 1 capsule)
  Interventions: Other: Ethyl Ester Marine Oil

INTERVENTIONS:
Other: Wax Ester Marine Oil — Wax ester marine oil (Calanus oil; 4 g providing 260 mg EPA and 156 mg DHA; 8 capsules) consumed once, in clinic, at t=0.
  Other Names: Calanus Oil; marine copepod Calanus finmarchicus
  Arms: Wax Ester Marine Oil
Other: Ethyl Ester Marine Oil — Ethyl ester (EE) marine oil (Lovaza OM3 EE; 1 g providing 465 mg EPA and 375 mg DHA; 1 capsule), consumed once, in clinic, at t=0
  Other Names: Lovaza
  Arms: Ethyl Ester Marine Oil

SUMMARY:
The objective of this study was to evaluate and compare the acute bioavailability of EPA and DHA in wax ester form provided as a dietary supplement compared to a well-studied and defined ethyl ester formulation in generally healthy men and women.

DETAILED DESCRIPTION:
A randomized, controlled two-period crossover study included one screening/baseline visit (visit 1, day -7) with four test visits during Period I (visits 2, 3, 4, and 5; days 0, 1, 2, and 3) and four tests visits during Period II (visits 6, 7, 8, and 9; days 14, 15, 16, and 17) with at least a 7-d washout between test periods. Eighteen healthy adults with fasting TAG concentrations <200 mg/dL were randomly assigned to one of two treatment sequences: receive 8 capsules containing Calanus oil® (Calanus AS, Tromso, Norway) supplying a total of 4 g of oil providing 260 mg EPA and 156 mg/day DHA primarily as wax esters, followed by 1 capsule supplying 1 g of oil providing 465 mg EPA and 375 mg DHA as ethyl esters (Lovaza®, GlaxoSmithKline, Research Triangle Park, NC); or, to receive Lovaza followed by Calanus Oil. Product was dispensed in-clinic with an standardized EPA- and DHA- free breakfast meal (t=0). Blood samples were obtained in-clinic at t= -30 min, and 1, 2, 4, 6, 8, 10 and 12 h timepoints. Subjects were provided a standardized EPA- and DHA-free meal at t=4 h and t=8. Subject were dismissed from the clinic after t-12 h blood draw and returned the morning of days 1, 2 and 3 (days 15, 16 and 17) for a 24 h, 48 h and 72 h fasting blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-59 years of age, inclusive.
2. BMI of ≥18.50 and ≤29.99 kg/m2 at visit 1 (day -7).
3. Fasting TG <200 mg/dL at visit 1 (day -7).
4. Score of 7 to 10 on the Vein Access Scale at visit 1 (day -7).
5. No health conditions that would prevent the subject from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
6. Willing to refrain from consumption of all fish/seafood (including shellfish), and/or EPA- or DHA-containing foods and supplements 14 d prior to visit 2 (day 0) and throughout the study.
7. Willing to limit alcohol consumption to no more than 1 drink/d following visit 1 (day -7) and throughout the study.
8. Non-smoker with no plans to change smoking habits during the study period.
9. Willing to maintain habitual diet (with the exception of foods to be restricted), physical activity patterns, and body weight throughout the trial.
10. Understood the study procedures and signed forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Abnormal laboratory test results of clinical significance at visit 1 (day -7), at the discretion of the Investigator. One re-test was allowed on a separate day prior to visit 2 (day 0) for subjects with abnormal laboratory test results.
2. History or presence of clinically important endocrine (including type 1 or 2 diabetes mellitus), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric or biliary disorders.
3. History or presence of a GI disorder that, in the judgment of the Investigator, may have disrupted normal digestion and absorption of the study products.
4. History of difficulty swallowing tablets/capsules that could have affected ability to consume the study products.
5. Extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Investigator.
6. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at visit 1 (day -7). One re-test was allowed on a separate day prior to visit 2 (day 0), for subjects whose blood pressure exceeded either of these cut points, in the judgment of the Investigator.
7. History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
8. Weight loss or gain >4.5 kg in the 3 months prior to visit 1 (day -7).
9. Use of medications or dietary supplements known to alter lipid concentrations within 4 weeks of visit 1 (day -7). Dietary supplements included, but were not limited to, the following: sterol/stanol products; dietary fiber supplements (including >1 teaspoon Metamucil® or viscous fiber-containing supplement per day); red rice yeast supplements; garlic supplements; soy isoflavone supplements; or niacin or its analogues at dosages >50 mg/day (or others at the discretion of the Investigator).
10. Use of non-study related omega-3-acid ethyl ester drug(s) or dietary supplement(s) with ≥1.0 g/d of EPA, DHA, or a combination of EPA and DHA within 4 months of visit 1 (day -7).
11. Known allergy or sensitivity to omega-3 fatty acids, fish, other seafood, or any ingredient in the study product or study meals.
12. Active infection or use of antibiotics within 5 d of visits 2 and 6 (days 0 and 14). Subjects that had an active infection and/or were using antibiotics were required to wait at least 5 d after the infection resolved or antibiotic use was complete prior to the first day of each test period (visits 2 and 6, days 0 and 14).
13. Female who was pregnant, planning to be pregnant during the study period, lactating, or was of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception was recorded in the source documentation.
14. Exposure to any non-registered drug product within 30 d prior to visit 1 (day -7).
15. Recent history of (within 12 months of screening; visit 1, day -7) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC) for plasma EPA+DHA | pre-product consumption (t = -0.5 h) to 72 h (iAUC-0.5-72h)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) and time to Cmax (Tmax) for EPA, DHA, and EPA+DHA | pre-product consumption (t = -0.5 h) to 72 h
iAUCs for plasma EPA+DHA | pre-product consumption (t = -0.5 h) to 24 h (iAUC-0.5-24 h), and to 48 h (iAUC-0.5-48 h)
The iAUCs for plasma EPA and DHA alone | (iAUC-0.5-24 h, iAUC-0.5-48 h, iAUC-0.5-72 h).

CONTACTS AND LOCATIONS:
Overall Officials: Chad Cook, PhD, Study Director — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided